CLINICAL TRIAL: NCT03857776
Title: A Phase Two Parallel-group Randomized Controlled Trial Assessing the Efficacy of Open Dialogue About Complementary Alternative Medicine (CAM) Integrated in Conventional Oncology Care
Brief Title: Open Dialogue About Complementary Alternative Medicine (CAM) Integrated in Conventional Oncology Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CAMONCO
Record Dates: First submitted 2019-02-22; First posted 2019-02-28 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Cancer
Keywords: Randomized controlled trial; Neoplasm; Communication; Complementary medicine; Integrative care; Integrative medicine
MeSH Terms: conditions — Neoplasms; Communication | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open dialogue about CAM (Other): Participation in an open dialogue about CAM with a nurse specialist. The dialogue will be based on the fundamentals of person-centered care and include patient preferences and wishes, reliable information and counselling, and advice about the potential risks and benefits of using CAM.
  The dialogue is estimated to last approximately 60 minutes and all dialogues will be conducted by the same nurse. Depending on patient needs and wishes there may be a follow-up consultation one month after the first dialogue.
  Interventions: Other: Open dialogue about complementary alternative medicine
- Standard care (Other): Standard care including referral to a homepage about complementary alternative medicine
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Open dialogue about complementary alternative medicine — 1-hour dialogue about CAM with a nurse specialist as an Integrated part of conventional oncology care
  Arms: Open dialogue about CAM
Other: Standard care — Standard care including referral to a homepage about CAM
  Arms: Standard care

SUMMARY:
The purpose of this phase two parallel-group randomized controlled trial is to assess the efficacy of open dialogue about CAM integrated in conventional oncology care. The investigators hypothesize that patients in the intervention group participating in a scheduled open dialogue with a nurse specialist about CAM will experience better physical and mental health compared to patients in the control group receiving standard care alone.

DETAILED DESCRIPTION:
Patients randomized to the intervention group will participate in a scheduled open dialogue about CAM with a specialist nurse, who has completed the Fellowship in Integrative Medicine at the University of Arizona. This is a training program for health professionals in empowering individuals and communities to optimize health and well-being through evidence-based, sustainable and integrative approaches. The open dialogue will be based on the fundamentals of person-centered care according to this program and include patient preferences and wishes, reliable information and counselling and advice about the potential risks and benefits of using CAM as an adjunct to conventional oncology care.

All dialogue, each lasting approximately 60 minutes, will be conducted by the same nurse as soon as possible and at the latest two weeks after enrolment. According to patient needs and wishes there may be a follow-up dialogue over the telephone or in the Oncology Outpatient Clinic. The potential second dialogue is estimated to last approximately 30 minutes.

Participants in the control group will receive standard information including reference to www.KABcancer.dk, which is a website presenting research on CAM, including information about its potential effects and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or more
* Speaks and reads Danish
* Diagnosed with a new primary cancer or a relapse of cancer within the last 3 months
* Planned or initiated medical oncology treatment at the Department of Oncology, Vejle Hospital
* At least two months of oncology treatment is realistic based on clinical assessment
* Life expectancy of at least six months
* Informed consent

Exclusion Criteria:

-Participation in other trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2020-05-24 (Actual); Study Completion 2020-05-24 (Actual)

PRIMARY OUTCOMES:
Difference in frequency of adverse events grade 3-4 between the two arms | 8 weeks after enrolment
  Adverse events are graded according to the Common Terminology Criteria for Adverse Events (CTCAEv5)

SECONDARY OUTCOMES:
Difference in patient reported quality of life between the two arms | At baseline and after 12 and 24 weeks
  Quality of life will be measured using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ C30). The EORTC is composed of both multi item scales and single item measures. These include five functional scales, three symptom scales, a global health status and six single items. All of the scales and single items measures range in score from 0 to 100. A high score for functional scale represents a high/health level of functioning. A high score for the global health status represents a high quality of life. A high score for a symptom scale represents a high level of symptomatology/problems
Difference in patients' evaluation of received information between the two arms | At baseline and after 12 and 24 weeks
  Evaluation of received information will be measured using the European Organization for Research and Treatment of Cancer Quality of Life Information Questionnaire (EORTC QLQ-INFO25).
Difference in patient reported degree of anxiety and depression between the two arms | At baseline and after 12 and 24 weeks
  Anxiety and depression will be measured using the Hospital Anxiety and Depression Scale (HADS)
Difference in frequency of adverse events grade 3-4 between the two arms | At baseline and after 12 and 24 weeks
  Frequency of adverse events grade 3-4 will be measured by using Common Terminology Criteria for Adverse Events (CTCAEv5)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Henrik Jensen, Study Chair — Department of Oncology, Vejle Hospital
Locations (1):
- Vejle Hospital, Vejle, Denmark

IPD SHARING:
Plan to Share IPD: No